CLINICAL TRIAL: NCT01017549
Title: Post Market Clinical Study to Evaluate the Safety and Performance of the Axxent® Electronic Brachytherapy System in Women With Resected, Early Stage Breast Cancer
Brief Title: Post Market Study Using the Xoft Axxent System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xoft, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-04
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: Stage I; Stage II; Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Radiotherapy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): This is a single arm study where all patients are treated with FDA cleared electronic brachytherapy treatment.
  Interventions: Radiation: Electronic brachytherapy (Axxent System)

INTERVENTIONS:
Radiation: Electronic brachytherapy (Axxent System) — 3.4 Gy per fraction for 10 fractions for a total of 34 Gy.
  Other Names: Radiation therapy, Axxent, Xoft, eBx, EBT, brachytherapy

SUMMARY:
The purpose of this multi-center clinical study is to compile post market performance and safety data on the Axxent System.

DETAILED DESCRIPTION:
The purpose of this multi-center clinical study is to compile post market performance and safety data on the Axxent System for the delivery of radiation therapy as part of breast conserving therapy in women with resected, early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Tumor with Tis, T1, N0, M0 - (AJC Classification)
* Invasive ductal carcinoma or ductal carcinoma in situ
* Negative microscopic surgical margins of at least 1mm in all directions
* Adequate skin spacing between balloon surface and surface of the skin - (> 7mm)

Exclusion Criteria:

* Pregnancy or breast-feeding - (During the treatment portion of the study, sexually active women of childbearing age will be asked to use pregnancy prevention)
* Scleroderma, systemic sclerosis and active lupus
* Infiltrating lobular histology

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-03-26 (Actual); Primary Completion 2013-06-06 (Actual); Study Completion 2016-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek K Mehta, MD, Principal Investigator — Swedish Cancer Institute
Locations (10):
- United States (10):
  - Mills Peninsula Hospital, San Mateo, California
  - Wellstar-Kennestone Cancer Center, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Holy Cross Medical Center, Silver Spring, Maryland
  - Beth Israel Medical Center, New York, New York
  - Dickstein Cancer Center- White Plains Hospital, White Plains, New York
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mehta VK, Algan O, Griem KL, Dickler A, Haile K, Wazer DE, Stevens RE, Chadha M, Kurtzman S, Modin SD, Dowlatshahi K, Elliott KW, Rusch TW. Experience with an electronic brachytherapy technique for intracavitary accelerated partial breast irradiation. Am J Clin Oncol. 2010 Aug;33(4):327-35. doi: 10.1097/COC.0b013e3181d79d9e. PMID 20375833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals with radiation oncology departments who had acquired the Xoft Axxent system and were qualified to be in the study were chosen as the 10 sites. Breast surgeons and radiation oncologists were the site investigators at 10 sites.
Pre-assignment Details: This was a single arm study, no randomization. Some patients consented but fell out of the study due to not meeting all eligibility (I/E) criteria after consenting to participation. 61 patients provided consent, 44 were treated.
Groups:
- Electronic Brachytherapy: Radiation therapy was delivered using the 510(k) cleared Xoft Axxent System. Accelerated partial breast irradiation is the method of radiation therapy administration that has been commonly used by physicians using Iridium-192, but was FDA cleared for use prior to commencing study enrollment using an electronic source.
Period: Eligibility Through 6 Month Follow-up
Arm/Group | Electronic Brachytherapy
Started | 44
Completed | 43 (6 month follow-up complete Oct 2008; data through 6 months and 1 year are published.)
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: One-year Follow-up
Arm/Group | Electronic Brachytherapy
Started | 43
Completed | 36
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 5
Period: 5 Year Follow-up
Arm/Group | Electronic Brachytherapy
Started | 36
Completed | 24
Not Completed | 12
Not completed — Lost to Follow-up | 9
Not completed — Mastectomy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Electronic Brachytherapy
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.24)
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 50 years | 2
  >=50 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delivery of 34 Gy in 10 Fractions
Description: Successful delivery of the radiation treatment defined as a total 34 Gy in a total of 10 fractions, 3.4 Gy per fraction. (Gray = GY is a measure of radiation dose delivered to tissue)
Time Frame: measured at end of 10th fraction, usually within 7 days
Population: All patients treated were analyzed
Measure: Number; unit: Participants
Arm/Group | Electronic Brachytherapy
Number analyzed (Participants) | 44
Participants | 42

2. Secondary Outcome: Serious Adverse Device Related Events Reported During the Course of the Study Through 6 Month Follow-up.
Description: Serious adverse device related events reported from treatment through 6 month follow-up and at 5-year follow-up are reported.
Time Frame: Through 6 months
Population: All patients treated were analyzed at 6 months except for 1 patient who was lost to follow-up.
Measure: Number; unit: events
Arm/Group | Electronic Brachytherapy
Number analyzed (Participants) | 44
events | 0

ADVERSE EVENTS:
Time Frame: Treatment through 5 Year Follow-up.
Description: Common Terminology Criteria V3 was used to report Adverse Events in this study.
Arm/Group | Electronic Brachytherapy
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 22/44
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Brachytherapy (N=44)
Erythema (Skin and subcutaneous tissue disorders) | 8 (8) — Erythema grade 2
Pain (Reproductive system and breast disorders) | 5 (5) — Pain CTC grade 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3) — Hyperpigmentation grade 2
Moist desquamation (Skin and subcutaneous tissue disorders) | 2 (2) — Moist desquamation grade 3
Infection (Infections and infestations) | 5 (5)
Seroma (Skin and subcutaneous tissue disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results are published; therefore the disclosure agreement is no longer in effect. The site investigators were to ask permission to publish single center results if they chose to publish prior to the entire study results were published.